CLINICAL TRIAL: NCT04499781
Title: Adherence Connection for Counseling, Education, and Support (ACCESS) II
Acronym: ACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Jacobi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-01135
Record Dates: First submitted 2020-07-29; First posted 2020-08-05 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: The ACCESS II RCT uses a two group, parallel, longitudinal study design. Participants will be randomized to the ACCESS synchronous peer intervention or the asynchronous web-based HIV ART adherence control. Block randomization will be used; the randomization scheme will be developed by the biostatistician and implemented in Research Electronic Data Capture (REDCap) to ensure that assignment to treatment condition is evenly distributed within each site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV-infected youth: Intervention (Experimental): Sample population of perinatally and behaviorally, HIV-infected youth (ages 18-29 years).
  Characteristics of the target study population include ethnic minority, Black and Hispanic HIV+AYA; both males and females are eligible for participation.
  Interventions: Behavioral: ACCESS II mHealth Intervention
- HIV-infected youth: control (Active Comparator): Sample population of perinatally and behaviorally, HIV-infected youth (ages 18-29 years).
  Characteristics of the target study population include ethnic minority, Black and Hispanic HIV+AYA; both males and females are eligible for participation.
  Interventions: Behavioral: ACCESS II control condition

INTERVENTIONS:
Behavioral: ACCESS II mHealth Intervention — Participants in the intervention condition will use videoconferencing to connect synchronously with trained HIV+ peer health coaches who will deliver eight weekly, 60-minute cognitive behavioral, motivational sessions for improved ART adherence.
  Arms: HIV-infected youth: Intervention
Behavioral: ACCESS II control condition — Web-based HIV adherence education. Participants in the control group will connect asynchronously to a web-based HIV ART adherence education condition.
  Arms: HIV-infected youth: control

SUMMARY:
The primary objective of the proposed clinical trial, Adherence Connection for Counseling, Education, and Support (ACCESS)-II, is to test the efficacy of ACCESS-II on antiretroviral treatment (ART) adherence and HIV-viral load in Black and Hispanic HIV-infected (HIV+) adolescents and young adults (AYA), ages 18-29 years (N=120) using a longitudinal (12 and 24 week outcomes), two-group, randomized control trial (RCT). Participants in the intervention condition will use videoconferencing to connect synchronously with trained HIV+ peer health coaches who will deliver eight weekly, 60-minute cognitive behavioral/motivational sessions for improved ART adherence. Participants in the control will connect asynchronously to a web-based HIV ART adherence education condition.

DETAILED DESCRIPTION:
To achieve these aims, a longitudinal (12 and 24- week study outcomes), two-group, randomized control trial (RCT) is proposed in a sample population of 120 perinatally and behaviorally, HIV-infected youth (ages 18-29 years). Participants in the intervention condition will use videoconferencing to connect synchronously with trained HIV+ peer health coaches who will deliver eight weekly, 60-minute cognitive behavioral47-50 motivational18 sessions for improved ART adherence. Participants in the control will connect asynchronously to a web-based HIV ART adherence education condition.

Study participants will access the intervention and control conditions outside of the clinical setting using study funded smart phones. Self-reported adherence and viral load (extracted from the medical records) of study participants will be measured, and uploaded to RedCAP. ART knowledge, adherence self-efficacy, HIV stigma, social support, psychological distress, and substance use will be measured using survey measures. Statistical analyses will be computed to assess the potential impact of ACCESS on adherence and HIV viral suppression, and will also be computed to assess changes in ART knowledge, adherence self-efficacy, HIV stigma, social support, psychological distress, and substance use among participants in both the intervention and control conditions.

ELIGIBILITY:
Inclusion criteria for participation in this study are:

* HIV seropositive status (perinatally and behaviorally infected youth)
* Ages 18-29 years
* English speaking
* Currently being prescribed an antiretroviral treatment regimen
* Evidence of virologic failure or (detectable quantitative HIV serum viral load>200 copies/ml)
* No neuro-cognitive deficits which would impede participation in videoconferencing sessions or completion of study measures

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Margaret Navarra, PhD, CPNP-PC, Principal Investigator — NYU Meyers College of Nursing
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to amd363@nyu.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements
Access Criteria: Requests may be directed to amd363@nyu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- ACCESS II mHealth Intervention: Sample population of perinatally and behaviorally, HIV-infected youth (ages 18-29 years).
  Characteristics of the target study population include ethnic minority, Black and Hispanic HIV+AYA; both males and females are eligible for participation.
  ACCESS II mHealth Intervention: Participants in the intervention condition will use videoconferencing to connect synchronously with trained HIV+ peer health coaches who will deliver eight weekly, 60-minute cognitive behavioral, motivational sessions for improved ART adherence.
- Control: Sample population of perinatally and behaviorally, HIV-infected youth (ages 18-29 years).
  Characteristics of the target study population include ethnic minority, Black and Hispanic HIV+AYA; both males and females are eligible for participation.
  ACCESS II control condition: Web-based HIV adherence education. Participants in the control group will connect asynchronously to a web-based HIV ART adherence education condition.
Period: Overall Study
Arm/Group | ACCESS II mHealth Intervention | Control
Started | 30 | 30
Completed | 26 | 27
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACCESS II mHealth Intervention | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (3.51) | 24.9 (2.9) | 24.95 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 14 | 15 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 13 | 26
  Not Hispanic or Latino | 17 | 17 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 18 | 37
  White | 2 | 0 | 2
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Self-Reported ART Adherence
Description: 3-day self-report of ART adherence was collected to describe subjective adherence behavior. Investigators will compute an cumulative average missed dose calculation: # of doses missed divided by total number of prescribed doses over the past 3 days. (scores range from 0 to 100%; higher scores = better adherence)
Time Frame: Baseline
Measure: Number; unit: Percentage of successful doses
Units Other Than Participants: Doses
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 30 | 30
Number analyzed (Doses) | 90 | 90
Percentage of successful doses | 56.67 | 58.7

2. Primary Outcome: Self-Reported ART Adherence
Description: as for outcome 1
Time Frame: Week 12
Population: 24 participants in the intervention arm were analyzed, as 2 withdrew from the study, 2 did not complete week-12 study activities and 2 were lost to follow-up.
Measure: Number; unit: Percentage of successful doses
Units Other Than Participants: Doses
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 24 | 30
Number analyzed (Doses) | 72 | 90
Percentage of successful doses | 74.64 | 71.79

3. Primary Outcome: Self-Reported ART Adherence
Description: 3-day self-report of ART adherence will be collected to describe subjective adherence behavior. Investigators will compute an average missed dose calculation: # of doses missed divided by total number of prescribed doses over the past 3 days. (scores range from 0 to 100%; higher scores = better adherence )
Time Frame: Week 24
Population: 26 participants in the intervention arm were analyzed, as 2 withdrew from the study and 2 were lost to follow-up. 27 participants in the control arm were analyzed, as 3 were lost to follow-up.
Measure: Number; unit: Percentage of successful doses
Units Other Than Participants: Doses
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 26 | 27
Number analyzed (Doses) | 78 | 81
Percentage of successful doses | 76.77 | 80.33

4. Primary Outcome: Log10 Viral Load
Description: Measured to eliminate the potential for social desirability bias associated with self-reported adherence. Viral load data was extracted from the medical records of participants.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Log10 Viral Load (Copies/mL)
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 30 | 30
Log10 Viral Load (Copies/mL) | 3.50 (1.2) | 3.40 (1.4)

5. Primary Outcome: Annualized Change in Log10 Viral Load (Copies/mL)
Description: Annualized change in log10 viral load is a useful metric for conveying change over time while accounting for varying time points and number of viral load data measurements. All available viral load data for study participants was included and some participants had more than 3 viral loads included.
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: log10 copies/mL/year
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 26 | 27
log10 copies/mL/year | -0.43 [-1.15 to 0.28] | -0.53 [-1.14 to 0.08]

6. Primary Outcome: Adherence Self-Efficacy Measured by the HIV Medication Taking Self-Efficacy Scale (HIV MT SES)
Description: Assessment of adherence self-efficacy. The HIV MT SES is a 26-item survey measure that uses an 10-point Likert scale (1=not confident; 10=completely confident) to assess HIV-medication taking self-efficacy belief and outcome expectancy. Higher scores indicate higher levels of self-efficacy.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 6.8 (2.0) | 6.8 (1.2)

7. Primary Outcome: Adherence Self-Efficacy Measured by the HIV Medication Taking Self-Efficacy Scale (HIV MT SES)
Description: as for outcome 6
Time Frame: Week 12
Population: 24 participants in the intervention arm were analyzed, as 2 withdrew from the study, 2 did not complete week-24 study activities and 2 were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 24 | 30
score on a scale | 8.0 (1.4) | 7.6 (1.2)

8. Primary Outcome: Adherence Self-Efficacy Measured by the HIV Medication Taking Self-Efficacy Scale (HIV MT SES)
Description: as for outcome 6
Time Frame: Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 26 | 27
score on a scale | 7.7 (1.6) | 7.4 (1.3)

9. Secondary Outcome: Knowledge About ART Measured With the HIV Treatment Knowledge Scale
Description: The HIV Treatment Knowledge Scale is a 21-item instrument that uses true and false questions to assess knowledge of adherence, side effects and antiretroviral resistance. The score is calculated as the number of correct responses; scores range from 0-21, where higher scores = increased knowledge.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 14.8 (3.1) | 14.5 (3.2)

10. Secondary Outcome: Knowledge About ART Measured With the HIV Treatment Knowledge Scale
Description: as for outcome 9
Time Frame: Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 24 | 30
score on a scale | 14.4 (3.8) | 14.8 (3.3)

11. Secondary Outcome: Knowledge About ART Measured With the HIV Treatment Knowledge Scale
Description: as for outcome 9
Time Frame: Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 26 | 27
score on a scale | 15.5 (3.4) | 15.8 (3.3)

12. Secondary Outcome: HIV Stigma Measured With the HIV Stigma Scale
Description: The HIV Stigma Scale is a 40-item questionnaire assessing HIV stigma. Each item is rated on a 4-point Likert scale ranging from 1-4. The total score is the sum of responses and ranges from 40 to 160; higher scores indicate a greater level of perceived HIV-related stigma.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 100.1 (21.1) | 105.9 (17.5)

13. Secondary Outcome: HIV Stigma Measured With the HIV Stigma Scale
Description: as for outcome 12
Time Frame: Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 24 | 30
score on a scale | 97.9 (18.9) | 103.3 (17.8)

14. Secondary Outcome: HIV Stigma Measured With the HIV Stigma Scale
Description: as for outcome 12
Time Frame: Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 26 | 27
score on a scale | 96.9 (21.4) | 101.4 (15.6)

15. Secondary Outcome: Depression Measured With the Patient Health Questionnaire-9 (PHQ-9)
Description: Depression was measured with the Patient Health Questionnaire (PHQ-9). The PHQ-9 includes 9 items from the DSM-IV criteria for depression with scores on a 4-point Likert scale (0=not at all, 3=nearly every day). The total score is the sum of responses and ranges from 0 to 27; higher scores indicate greater levels of depression.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 5.6 (6.3) | 7.7 (6.2)

16. Secondary Outcome: Depression Measured With the Patient Health Questionnaire-9 (PHQ-9)
Description: as for outcome 15
Time Frame: Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 24 | 30
score on a scale | 4.3 (5.0) | 5.6 (5.5)

17. Secondary Outcome: Depression Measured With the Patient Health Questionnaire-9 (PHQ-9)
Description: as for outcome 15
Time Frame: Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 26 | 27
score on a scale | 4.7 (5.6) | 5.7 (5.1)

18. Secondary Outcome: Anxiety Measured With the Generalized Anxiety Disorder-7 (GAD-7)
Description: Generalized anxiety disorder (GAD) was assessed with the Generalized Anxiety Disorder-7 (GAD-7). The measure includes 7 items about symptoms in the past two weeks. Each item is rated on 4-point Likert scale from 0-3. The total score is the sum of responses and ranges from 0-21; higher scores indicate greater levels of anxiety.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 6.3 (5.8) | 7.3 (5.9)

19. Secondary Outcome: Anxiety Measured With the Generalized Anxiety Disorder-7 (GAD-7)
Description: as for outcome 18
Time Frame: Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 24 | 30
score on a scale | 4.5 (4.3) | 6.0 (5.6)

20. Secondary Outcome: Anxiety Measured With the Generalized Anxiety Disorder-7 (GAD-7)
Description: as for outcome 18
Time Frame: Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 26 | 27
score on a scale | 5.0 (5.0) | 5.8 (5.4)

21. Secondary Outcome: Number of Participants With Trauma Measured With the Primary Care-PTSD Screen-5 (PC-PTSD)
Description: Post-traumatic stress disorder (PTSD) was measured with the Primary Care-PTSD Screen-5 (PC-PTSD). The PC-PTSD is a brief measure using four-items to screen for symptoms of PTSD (re-experiencing, numbness, hyperarousal and avoidance behaviors) in primary care or ambulatory settings. The total score is the number of "Yes" responses and ranges from 0-5. Higher scores indicate probable or positive screen for PTSD. A participant was considered to have "trauma" if they reported 3 or more trauma symptoms in the past month.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 30 | 30
Participants | 11 | 11

22. Secondary Outcome: Number of Participants With Trauma Measured With the Primary Care-PTSD Screen-5 (PC-PTSD)
Description: as for outcome 21
Time Frame: Week 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 24 | 30
Participants | 5 | 10

23. Secondary Outcome: Number of Participants With Trauma Measured With the Primary Care-PTSD Screen-5 (PC-PTSD)
Description: as for outcome 21
Time Frame: Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 26 | 27
Participants | 4 | 4

24. Secondary Outcome: Social Support and Isolation Measured With the Adolescent Medicine Trials Network (ATN) iTech Short Measure of the Patient-Reported Outcomes Measure Information System (PROMIS) Social Relationship Scales - Companionship Score
Description: The ATN short measure is a 20-item tool where each item is rated on a 5-point Likert scale (1-5). The Companionship subscale comprises 4 items of the ATN short measure. The subscale raw score is the sum of responses; the raw score is converted to a T-score ranging from 25.2-63.1 with a mean of 50 and standard deviation of 10; higher scores reflect greater companionship.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 30 | 30
T-score | 47.0 (2.7) | 46.9 (2.5)

25. Secondary Outcome: Social Support and Isolation Measured With the Adolescent Medicine Trials Network (ATN) iTech Short Measure of the Patient-Reported Outcomes Measure Information System (PROMIS) Social Relationship Scales - Companionship Score
Description: as for outcome 24
Time Frame: Week 12
Population: as for outcome 7
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 24 | 30
T-score | 50.1 (2.8) | 48.9 (2.8)

26. Secondary Outcome: Social Support and Isolation Measured With the Adolescent Medicine Trials Network (ATN) iTech Short Measure of the Patient-Reported Outcomes Measure Information System (PROMIS) Social Relationship Scales - Companionship Score
Description: as for outcome 24
Time Frame: Week 24
Population: as for outcome 3
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 26 | 27
T-score | 49.4 (2.8) | 48.0 (2.7)

27. Secondary Outcome: Social Support and Isolation Measured With the ATN iTech Short Measure of the PROMIS Social Relationship Scales - Emotional Support Score
Description: The ATN short measure is a 20-item where each item is rated on a 5-point Likert scale (1-5). The Emotional Support subscale comprises 4 items of the ATN short measure. The subscale raw score is the sum of responses; the raw score is converted to a T-score ranging from 25.7-62.0 with a mean of 50 and standard deviation of 10; higher scores reflect greater emotional support.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 30 | 30
T-score | 47.2 (2.8) | 46.7 (2.8)

28. Secondary Outcome: Social Support and Isolation Measured With the ATN iTech Short Measure of the PROMIS Social Relationship Scales - Emotional Support Score
Description: as for outcome 27
Time Frame: Week 12
Population: as for outcome 7
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 24 | 30
T-score | 48.5 (2.7) | 47.9 (2.7)

29. Secondary Outcome: Social Support and Isolation Measured With the ATN iTech Short Measure of the PROMIS Social Relationship Scales - Emotional Support Score
Description: as for outcome 27
Time Frame: Week 24
Population: as for outcome 3
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 26 | 27
T-score | 47.9 (2.8) | 46.7 (2.6)

30. Secondary Outcome: Social Support and Isolation Measured With the ATN iTech Short Measure of the PROMIS Social Relationship Scales - Informational Support Score
Description: The ATN short measure is a 20-item where each item is rated on a 5-point Likert scale (1-5). The Informational Support subscale comprises 4 items of the ATN short measure. The subscale raw score is the sum of responses; the raw score is converted to a T-score ranging from 25.6-65.6 with a mean of 50 and standard deviation of 10; higher scores reflect greater informational support.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 30 | 30
T-score | 47.1 (2.7) | 47.7 (2.7)

31. Secondary Outcome: Social Support and Isolation Measured With the ATN iTech Short Measure of the PROMIS Social Relationship Scales - Informational Support Score
Description: as for outcome 30
Time Frame: Week 12
Population: as for outcome 7
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 24 | 30
T-score | 51.3 (2.8) | 50.2 (3.0)

32. Secondary Outcome: Social Support and Isolation Measured With the ATN iTech Short Measure of the PROMIS Social Relationship Scales - Informational Support Score
Description: as for outcome 30
Time Frame: Week 24
Population: as for outcome 3
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 26 | 27
T-score | 51.3 (2.8) | 49.3 (2.8)

33. Secondary Outcome: Social Support and Isolation Measured With the ATN iTech Short Measure of the PROMIS Social Relationship Scales - Instrumental Support Score
Description: The ATN short measure is a 20-item where each item is rated on a 5-point Likert scale (1-5). The Instrumental Support subscale comprises 4 items of the ATN short measure. The subscale raw score is the sum of responses; the raw score is converted to a T-score ranging from 29.3-63.3 with a mean of 50 and standard deviation of 10; higher scores reflect greater instrumental support.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 30 | 30
T-score | 45.9 (2.8) | 44.0 (2.7)

34. Secondary Outcome: Social Support and Isolation Measured With the ATN iTech Short Measure of the PROMIS Social Relationship Scales - Instrumental Support Score
Description: as for outcome 33
Time Frame: Week 12
Population: as for outcome 7
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 24 | 30
T-score | 48.7 (3.0) | 47.3 (3.0)

35. Secondary Outcome: Social Support and Isolation Measured With the ATN iTech Short Measure of the PROMIS Social Relationship Scales - Instrumental Support Score
Description: as for outcome 33
Time Frame: Week 24
Population: as for outcome 3
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 26 | 27
T-score | 49.6 (3.0) | 48.8 (3.0)

36. Secondary Outcome: Social Support and Isolation Measured With the ATN iTech Short Measure of the PROMIS Social Relationship Scales - Social Isolation Score
Description: The ATN short measure is a 20-item where each item is rated on a 5-point Likert scale (1-5). The Social Isolation subscale comprises 4 items of the ATN short measure. The subscale raw score is the sum of responses; the raw score is converted to a T-score ranging from 34.8-74.2 with a mean of 50 and standard deviation of 10; higher scores reflect greater social isolation.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 30 | 30
T-score | 54.6 (2.9) | 56.3 (2.8)

37. Secondary Outcome: Social Support and Isolation Measured With the ATN iTech Short Measure of the PROMIS Social Relationship Scales - Social Isolation Score
Description: as for outcome 36
Time Frame: Week 12
Population: as for outcome 7
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 24 | 30
T-score | 50.7 (3.3) | 52.0 (2.9)

38. Secondary Outcome: Social Support and Isolation Measured With the ATN iTech Short Measure of the PROMIS Social Relationship Scales - Social Isolation Score
Description: as for outcome 36
Time Frame: Week 24
Population: as for outcome 3
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 26 | 27
T-score | 52.5 (3.3) | 52.7 (2.9)

39. Secondary Outcome: Tobacco - Lifetime Use
Description: Substance use was assessed with a modified Adolescent Trials Network (ATN) measure designed for use in clinical settings. Presented as the number of participants with lifetime tobacco use.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 30 | 30
Participants | 20 | 20

40. Secondary Outcome: Marijuana - Lifetime Use
Description: Substance use was assessed with a modified Adolescent Trials Network (ATN) measure designed for use in clinical settings. Presented as the number of participants with lifetime marijuana use.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 30 | 30
Participants | 23 | 25

41. Secondary Outcome: Alcohol - Lifetime Use
Description: Substance use was assessed with a modified Adolescent Trials Network (ATN) measure designed for use in clinical settings. Presented as the number of participants with lifetime alcohol use.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ACCESS II mHealth Intervention | Control
Number analyzed (Participants) | 30 | 30
Participants | 25 | 27

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Adverse event data were collected at baseline, 12 weeks, and 24 weeks study visit through standard questionnaire, PHQ-9 question #9, "Over the last 2 weeks, how often have you been bothered by any of the following problems? Thoughts that you would be better off dead, or of hurting yourself." Additionally, self-reporting by participants were also documented.
Arm/Group | ACCESS II mHealth Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 8/30 | 5/30
Other Adverse Events (participants affected / at risk) | 3/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACCESS II mHealth Intervention (N=30) | Control (N=30)
Self-report of injury from being stabbed (Injury, poisoning and procedural complications) | 0 | 1
Pneumocystis carinii pneumonia (PCP) and esophageal candidiasis (Infections and infestations) | 0 | 1
Self-report of suicidal thoughts within the past 2 weeks (Psychiatric disorders) | 6 | 2
Pneumonia (Infections and infestations) | 2 | 0
Self-report of hospitalization for kidney stones (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACCESS II mHealth Intervention (N=30) | Control (N=30)
Self-report of nervous breakdown, "not doing well mentally, physically, emotionally" (Psychiatric disorders) | 1 | 0
Self-reported incarceration (Social circumstances) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT04499781/Prot_SAP_000.pdf